CLINICAL TRIAL: NCT00941954
Title: Walking Away From Type 2 Diabetes: a Cluster Randomized Controlled Trial to Investigate the Effect of Structured Education on Walking Activity in Those With a High Risk of Developing Type 2 Diabetes
Brief Title: Walking Away: Structured Education Versus Written Information for Individuals With High Risk of Developing Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: University of Leicester (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LNR CLRN 10343
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes
Keywords: Physical activity; Diabetes; Prevention; Pedometer; Walking; Structured education; Randomized; Risk score; Impaired glucose regulation
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental): A group-based structured educational programme.
  Interventions: Behavioral: Structured Education
- Control (Active Comparator): Written Information (booklet).
  Interventions: Behavioral: Written Information

INTERVENTIONS:
Behavioral: Structured Education — The intervention group will be offered a group-based structured educational programme aimed at promoting increased ambulatory activity by targeting perceptions and knowledge of diabetes risk, physical activity self-efficacy, barriers to physical activity and self-regulatory skills based on pedometer use. The programme will employ a person-centred approach to patient education that is based on self-management programmes for individuals with type 2 diabetes and prediabetes that have been developed and tested by our research group. The programme will be designed to be delivered to 5-10 participants by two trained educators and is 3.5 hours long. Brief follow-up counselling will be offered once every 6 months.
  Arms: Lifestyle counseling
Behavioral: Written Information — Control subjects will receive a booklet detailing information on risk factors for type 2 diabetes (T2DM) and cardiovascular disease (CVD) and how physical activity can be used to prevent T2DM and CVD.
  Arms: Control

SUMMARY:
Diabetes is a debilitating chronic disease reaching epidemic proportions. Lack of physical activity is a key factor driving this epidemic and it is therefore vital that workable methods of encouraging people to exercise and reducing inactivity are developed and tested if we are to stem the rising tide of diabetes.

This cluster randomised controlled trial will investigate whether a person-centred group educational programme can increase walking activity and reduce the risk of developing diabetes in high-risk individuals identified in primary care settings. In total 804 patients will be recruited to the study. Physical activity levels, glucose control, incidence of type 2 diabetes and anthropometric measurements (e.g. weight) will be tested on an annual basis over three years.

This trial will be the first to test the feasibility, efficacy and value for money of a physical activity intervention aimed at reducing the risk of diabetes in a community setting in a multi-ethnic population in the UK.

Primary research hypothesis: A pragmatic structured education programme aimed at promoting walking activity initiates long-term increases in physical activity in individuals identified through a risk score as having an increased risk of developing type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 18+
* High risk of developing type 2 diabetes as identified through a risk score

Exclusion Criteria:

* Diagnosed diabetes
* Taking steroid medication
* Serious chronic illness preventing participation in trial
* Unable to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2009-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in ambulatory activity (walking) | 12 months

SECONDARY OUTCOMES:
Light-, moderate- and vigorous-intensity physical activity | 12 months; 24 months; 36 months
Time spent in sedentary activities | 12 months; 24 months; 36 months
Fasting and 2-hour post-challenge plasma glucose | 12 months; 24 months; 36 months
Glycosylated hemoglobin (HbA1c) | 12 months; 24 months; 36 months
Advanced glycation end products | 12 months; 24 months; 36 months
Fasting and 2-hour post-challange plasma insulin | 12 months; 24 months; 36 months
Adipokines (leptin, interleukin 6 and tumor necrosis factor alpha) | 12 months; 24 months; 36 months
C-reactive protein | 12 months; 24 months; 36 months
Standard anthropometric variables | 12 months; 24 months; 36 months
Visceral adiposity (sub-set of participants) | 12 months; 24 months; 36 months
Muscle mass (sub-set of participants) | 12 months; 24 months; 36 months
Illness perceptions and efficacy beliefs | 12 months; 24 months; 36 months
Health related quality of life | 12 months; 24 months; 36 months
Depression | 12 months; 24 months; 36 months
Change in ambulatory activity (walking) | 24 months; 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J Davies, MD, Principal Investigator — University of Leicester; University Hospitals of Leicester NHS Trust
Locations (1):
- University Hospitals of Leicester (UHL), Leicester, United Kingdom

REFERENCES:
- [Derived] Yates T, Gray LJ, Henson J, Edwardson CL, Khunti K, Davies MJ. Impact of Depression and Anxiety on Change to Physical Activity Following a Pragmatic Diabetes Prevention Program Within Primary Care: Pooled Analysis From Two Randomized Controlled Trials. Diabetes Care. 2019 Oct;42(10):1847-1853. doi: 10.2337/dc19-0400. Epub 2019 Aug 9. PMID 31399440
- [Derived] Henson J, Edwardson CL, Morgan B, Horsfield MA, Khunti K, Davies MJ, Yates T. Sedentary Time and MRI-Derived Measures of Adiposity in Active Versus Inactive Individuals. Obesity (Silver Spring). 2018 Jan;26(1):29-36. doi: 10.1002/oby.22034. PMID 29265769
- [Derived] Bodicoat DH, O'Donovan G, Dalton AM, Gray LJ, Yates T, Edwardson C, Hill S, Webb DR, Khunti K, Davies MJ, Jones AP. The association between neighbourhood greenspace and type 2 diabetes in a large cross-sectional study. BMJ Open. 2014 Dec 23;4(12):e006076. doi: 10.1136/bmjopen-2014-006076. PMID 25537783
- [Derived] Yates T, Davies MJ, Henson J, Troughton J, Edwardson C, Gray LJ, Khunti K. Walking away from type 2 diabetes: trial protocol of a cluster randomised controlled trial evaluating a structured education programme in those at high risk of developing type 2 diabetes. BMC Fam Pract. 2012 May 29;13:46. doi: 10.1186/1471-2296-13-46. PMID 22642610